CLINICAL TRIAL: NCT07301723
Title: A Single-center, Open-label Trial to Determine the Absolute Bioavailability of Cenerimod Using an Intravenous 14C-radiolabeled Cenerimod Microtracer in Healthy Male Participants
Brief Title: A Trial to Evaluate the Absolute Bioavailability of Cenerimod in Healthy Male Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ID-064-108
Record Dates: First submitted 2025-11-17; First posted 2025-12-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — cenerimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cenerimod (Experimental): Cenerimod is administered as a single oral dose followed by a single i.v. radiolabeled dose 6 h later.
  Interventions: Drug: Cenerimod (oral); Drug: 14C-Cenerimod (i.v.)

INTERVENTIONS:
Drug: Cenerimod (oral) — A single dose of cenerimod, administered as an oral tablet at a strength of 4 mg
  Other Names: ACT-334441
Drug: 14C-Cenerimod (i.v.) — A single i.v. dose of 7.5 µg 14C-radiolabeled cenerimod (34.5 kBq), with administration starting 6 h after administration of the oral dose.
  Other Names: 14C-ACT-334441

SUMMARY:
The goal of this clinical trial is to learn about the absolute bioavailability of cenerimod in healthy participants. It will also provide information about the safety of cenerimod.

Participants will receive one tablet with cenerimod, followed by an intravenous (i.v.) infusion with a 14C-radiolabeled cenerimod microtracer (cenerimod with a very low dose of radioactivity) 6 hours later.

Participants will stay at the clinic for a total of 4 days, and will return to the clinic for further tests over the course of approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form in a language understandable to the participant prior to any trial-mandated procedure.
2. Healthy male participant aged between 18 and 65 years (inclusive) at Screening. Healthy is defined as no clinically relevant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs measurements, and clinical laboratory evaluations.
3. Body mass index 18.0-29.9 kg/m^2 (inclusive) at Screening.
4. Ability to communicate well with the investigator, in a language understandable to the participant, and to understand and comply with the trial requirements.
5. Systolic blood pressure 90-140 mmHg, diastolic blood pressure 60-90 mmHg, and pulse rate 55-100 bpm (inclusive), measured on either arm (same arm used for both Screening and on the day of study treatment administration), after 5 min in the supine position at Screening and prior to oral dosing on the day of study treatment administration.
6. 12-lead safety ECG: QTcF < 450 ms, QRS interval < 120 ms, PR interval < 200 ms, and heart rate 55-100 bpm, and without clinically relevant abnormalities, measured after 5 min in the supine position at Screening and prior to oral dosing on the day of study treatment administration.

Main Exclusion Criteria:

1. Previous exposure to cenerimod.
2. Known hypersensitivity to any excipients of the trial intervention formulations.
3. Known hypersensitivity or allergy to natural rubber latex.
4. History of major medical or surgical disorders which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the trial interventions (appendectomy and herniotomy allowed, cholecystectomy not allowed).
5. Acute, ongoing, recurrent, or chronic systemic disease able to interfere with the evaluation of the trial results.
6. Clinically relevant history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
7. Lymphopenia (< 0.9 x 10^9 cells/L) at Screening or on the day prior to study treatment administration.
8. Family history of sick-sinus syndrome.
9. Any cardiac condition or illness (including ECG abnormalities) with a potential to increase the cardiac risk of the participant based on the standard 12-lead ECG at Screening or pre-dose on the day of study treatment administration.
10. History or presence of cardiac rhythm disorders (e.g., sinoatrial heart block, sick-sinus syndrome, 2nd or 3rd degree atrioventricular block, long QT syndrome, symptomatic bradycardia, atrial flutter, or atrial fibrillation).
11. Previous treatment with antiarrhythmic medications of class Ia or III within 2 weeks or 5 elimination half-lives, whichever is longer, prior to oral dosing.
12. Clinically relevant findings in clinical laboratory tests (hematology, clinical chemistry, and urinalysis) at Screening or on the day prior to study treatment administration.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Absolute bioavailability | Up to 98 days post-dose
  Absolute bioavailability of a single oral dose of 4 mg cenerimod, calculated as: area under the plasma concentration-time curve from zero to infinity (AUC0-∞) of the oral dose / AUC0-∞ of the intravenous dose, normalized by dose.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (1):
- Pharmaceutical Research Associates Group B.V., Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No